CLINICAL TRIAL: NCT01443611
Title: The Relevance of Performing Lumbar Puncture in Infants Aged 3 to 12 Months With First Episode of Febrile Convulsion
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B and Pediatric Hematology Unit, HaEmek Medical Center, Israel
Other Study IDs: 0138-10-EMC
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Febrile Convulsions
Keywords: Infants
MeSH Terms: conditions — Seizures, Febrile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with first episode of Febrile Convlusions

SUMMARY:
The actual recommendations for infants aged 3 to 12 months presented with first episode of Febrile Convulsions highly recommend performing lumbar puncture in order to rule out Bacterial Meningitis. On the other hand, recent studies in the era of anti Pneumococcal vaccination arise the question if in the presence of a normal physical examination those recommendations are still relevant. The purpose of this study is to summarized retrospectively the clinical records of all the infants admitted to the pediatric wards in the ten years period since 2000 to 2010 in order to record the incidence of Bacterial Meningitis among infants admitted with the First episode of Febrile Convulsions.

DETAILED DESCRIPTION:
Demographic data, including ethnic origin, age an gender will be recorded. The type of Convulsions (Simple or Complex), duration, and time since the fever was noticed will be also recorded. Another data that will be summarized included: previous antibiotic treatment, physical examination with special emphasis on neurological examination and meningeal signs, routine laboratory analysis including blood count and cerebrospinal fluid (CSF) results and the final diagnosis including the cause of fever.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 3 to 12 months who presents with First Episode of Febrile Convulsions during the period 1/1/2000 until 31/12/2010

Exclusion Criteria:

* infants with previous neurological diseases, or
* recent neurological disease that are not included in the characteristics of Febrile Convulsion

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged 3 to 12 months who presents with First Episode of Febrile Convulsions
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal lumbar puncture | One year
  The number of patients aged six months to one year that underwent lumbar puncture when they were admitted with simple febrile convulsions

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Dpt B - Ha'Emek Medical Center, Afula, Afula, Israel